CLINICAL TRIAL: NCT01665638
Title: A Double-Blind, Randomized, Placebo-Controlled, 2-Way Cross-Over Study to Evaluate the Effect of Single Dose Canagliflozin on Kinetics of C-Peptide in Healthy Subjects
Brief Title: Effects of Canagliflozin on C-peptide Clearance in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: CR100800; 28431754DIA1049 (Other: Janssen-Cilag International NV); 2012-001667-73 (EudraCT Number)
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Healthy; Clearance; Canagliflozin; JNJ-28431754; Placebo; Somatostatin; C-peptide
MeSH Terms: interventions — Canagliflozin; Somatostatin; C-Peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence Group AB (Experimental)
  Interventions: Drug: Canagliflozin 300 mg; Drug: Placebo; Drug: Somatostatin; Drug: C-peptide
- Treatment Sequence Group BA (Experimental)
  Interventions: Drug: Canagliflozin 300 mg; Drug: Placebo; Drug: Somatostatin; Drug: C-peptide

INTERVENTIONS:
Drug: Canagliflozin 300 mg — Singe over-encapsulated 300 mg tablet of canagliflozin administered orally (by mouth) on Day 1 of Treatment Period 1 or Day 1 of Treatment Period 2.
Drug: Placebo — Singe capsule of placebo administered orally (by mouth) on Day 1 of Treatment Period 1 or Day 1 of Treatment Period 2.
Drug: Somatostatin — A primed (50 mcg in 1 mL sterile 0.9% NaCl solution i.v. injection over 1 minute) constant (500 mcg/hour) i.v. infusion of somatostatin for 4 hours approximately 2 hours after canagliflozin or placebo dosing on Day 1 of Treatment Period 1 and Day 1 of Treatment Period 2. The total dose of somatostatin administered during each period will be 50 mcg + 500 mcg/hour x 4 hours = 2050 mcg.
Drug: C-peptide — Single bolus dose of 150 mcg synthetic human C-peptide in 1 mL water for injection administered i.v. (in the vein) approximately 3 hours after canagliflozin or placebo dosing on Day 1 of Treatment Period 1 and Day 1 of Treatment Period 2.

SUMMARY:
The purpose of this study is to assess whether treatment with a single oral 300 mg dose of canagliflozin alters the kinetics (ie, clearance/removal from body) of serum C-peptide (a protein released from the pancreas during insulin secretion) in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a double-blind (neither the volunteer nor the study doctor/staff will know the identity of the assigned treatments) study to assess the effect of single oral (taken by mouth) dose of canagliflozin on clearance (removal from the body) of C-peptide in healthy adult volunteers. Healthy volunteers will be randomly (by chance) assigned to receive a single oral dose of canagliflozin followed by a single oral dose of placebo (inactive substance) or a single dose of placebo followed by a single dose of canagliflozin with a period of 7-10 days between treatments. Healthy volunteers will also receive intravenous (i.v.) infusion (injection in the vein) of somatostatin for 4 hours and a single dose i.v. injection of synthetic human C-peptide following administration of canagliflozin or placebo during each treatment period. Somatostatin will suppress the normal secretion of C-peptide, a protein that is released from the pancreas during insulin secretion, so that the human C-peptide administered to volunteers can be accurately measured. The total study duration for each volunteer will be approximately 44 days. During the study, blood and urine samples will be drawn (collected) for clinical laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 18 and 30 kg/m2, inclusive, and a body weight of not less than 50 kg

Exclusion Criteria:

* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy or clinically significant adverse reactions to canagliflozin or placebo or any of the excipients of the canagliflozin or placebo formulation
* Known hypersensitivity of synthetic human C-peptide, somatostatin preparation, or other structurally related peptides

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in C-peptide kinetic parameters | Before and after study drug administration on Day 1 of Treatment Periods 1 and 2
  Parameters are volume of distribution (Vd), clearance (CL) and half life (T1/2)

SECONDARY OUTCOMES:
The number of volunteers who report adverse events | Up to 22 days following Day 1 of Treatment Period 1

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Neuss, Germany